CLINICAL TRIAL: NCT01079429
Title: Large Scale Study of DNA Copy Numbers Variations and Gene Expression Profile of Bone Marrow Plasma Cells From Monoclonal Gammopathy of Undetermined Significance (MGUS) and Indolent Myeloma (SMM).
Brief Title: Study of DNA Copy Numbers Variations and Gene Expression Profile of Bone Marrow Plasma Cells From MGUS and SMM.
Acronym: GENOMGUS
Status: Terminated | Type: Observational
Why Stopped: sponsor and investigator 's decision
Sponsor: Rennes University Hospital (Other)
Collaborators: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Other Study IDs: RCB 2008-A01023-52; AFSSAPS B80894-60 (Other: AFSSAPS); IFM 08-02 (Other: IFM)
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Myeloma
Keywords: Monoclonal gammopathy of undetermined significance; MGUS; Smoldering myeloma; SMM; Multiple myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Plasma Urine Bone marrow
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MGUS or SMM: Patients with Monoclonal gammopathy of undetermined significance or smoldering myeloma
  Interventions: Genetic: Genetic study of DNA copies

INTERVENTIONS:
Genetic: Genetic study of DNA copies — Gene expression profiling, DNA copy number variation

SUMMARY:
The purpose of this study is to describe DNA copy number variations and gene expression profiles of bone marrow plasma cells of monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM). The final objective is to search for correlations with the risk of progression in order to establish a predictive model of early malignant transformation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 70 years
* Written informed consent
* One of the following three criteria:

  * Recently diagnosed IgG or IgA monoclonal gammopathy without clinical or biological features of malignant hemopathy
  * IgG or IgA MGUS regardless the date of the diagnosis
  * SMM regardless the date of the diagnosis
* Normal blood count, creatininemia and calcemia *
* Bence-Jones proteinuria below 1g/24 hours
* Absence of bone pain
* No clinical or biological features of amyloidosis
* No recurrent episode of infection (more than 2 infections requiring antibiotics in the previous 6 months) * In case of abnormal blood count, renal failure or hypercalcemia, patients may be included if an intercurrent cause is identified (for example anemia associated with iron deficiency)

Diagnostic criteria for MGUS:

* Monoclonal component concentration below 30 g / l AND
* Bone marrow plasmacytosis below 10%
* Bence-Jones proteinuria below 1g/24 hours
* Normal blood count, creatininemia and calcemia *
* Absence of bone lesions on conventional bone radiographies
* No clinical or biological features of amyloidosis
* Absence of hyperviscosity syndrome
* No recurrent episode of infection (more than 2 infections requiring antibiotics in the previous 6 months) * In case of abnormal blood count, renal failure or hypercalcemia, patients may be included if an intercurrent cause is identified (for example anemia associated with iron deficiency)

Diagnostic criteria for SMM:

* Monoclonal component concentration greater than 30 g / l AND / OR
* Bone marrow plasmacytosis greater than 10%
* Bence-Jones proteinuria below 1g/24 hours
* Normal blood count, creatininemia and calcemia *
* Absence of bone lesions on conventional bone radiographies
* No clinical or biological features of amyloidosis
* Absence of hyperviscosity syndrome
* No recurrent episode of infection (more than 2 infections requiring antibiotics in the previous 6 months) * In case of abnormal blood count, renal failure or hypercalcemia, patients may be included if an intercurrent cause is identified (for example anemia associated with iron deficiency)

Exclusion Criteria:

* Patients younger than 18 years
* Patients older than 71 years
* IgM monoclonal gammopathy (regardless of diagnosis)
* Monoclonal gammopathy associated with hematologic malignancies (multiple myeloma, chronic lymphocytic leukemia, ...)
* Patients with chronic liver disease, autoimmune or neoplastic disease for less than 5 years
* Active viral hepatitis B or C
* HIV seropositive patient
* Pregnant woman
* Breastfeeding woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Monoclonal gammopathy of undetermined significance or Smoldering myeloma
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2009-01-12 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Progression to symptomatic multiple myeloma | Every 6 or 12 months during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DECAUX, MD, Principal Investigator — Rennes University Hospital
Locations (27):
- France (27):
  - Rennes University Hospital, Rennes, Brittany Region
  - Nantes University Hospital, Nantes, Pays de Loire
  - CHU Amiens - médecine interne, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier H.Duffaut - Avignon, Avignon
  - Hôpital Jean Minjoz - Besancon, Besançon
  - Service de Médecine interne - Centre Hospitalier, Blois
  - Bordeaux Bergonié, Bordeaux
  - Bordeaux Haut Leveque, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital A.Morvan Brest, Brest
  - Centre F.Baclesse, Caen
  - CHU Caen, Caen
  - Hôpital d'instruction des armées Percy, Clamart
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CH Colmar, Colmar
  - CH Dijon, Dijon
  - CHG Dunkerque, Dunkirk
  - CH Grenoble, Grenoble
  - CH La Roche sur yon, La Roche-sur-Yon
  - CH Laval, Laval
  - Le Mans Victor Hugo, Le Mans
  - Hôpital Claude Huriez, Lille
  - Centre Hospitalier Yves Le Foll de Saint Brieuc - Service d'Hématologie, Saint-Brieuc
  - CHU Toulouse Purpan, Toulouse
  - CHU Toulouse Rangueil, Toulouse
  - Service d'Hématologie - Hôpital de Brabois, Vandœuvre-lès-Nancy